CLINICAL TRIAL: NCT03983538
Title: A Single Center Pilot Study Evaluating the Use of Mathematical Modeling to Predict Response to Neoadjuvant Anthracycline / Taxane Based Chemotherapy in Women With HER2 Negative Stage II and III Breast Cancer
Brief Title: Mathematical Modeling to Predict Response to Neoadjuvant Chemotherapy in Breast Cancer
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 1411
Record Dates: First submitted 2019-06-04; First posted 2019-06-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving chemotherapy: Patients receive a protocol-approved chemotherapy regimen containing Doxorubicin (or Epirubicin), Cyclophosphamide, and Paclitaxel (or Docetaxel) based on the patient and/or physician preference.
  Interventions: Other: Mathematical modeling to predict response to chemotherapy

INTERVENTIONS:
Other: Mathematical modeling to predict response to chemotherapy — Mathematical modeling using the patient's diagnostic core biopsy and baseline MRI of the breast will be used to predict the response to above therapy.

SUMMARY:
This is a feasibility study evaluating the use of a mathematical model to predict response to standard neoadjuvant anthracycline / taxane based chemotherapy in patients with breast cancer.

DETAILED DESCRIPTION:
This is a feasibility study evaluating the use of a mathematical model to predict response to standard neoadjuvant chemotherapy in patients with breast cancer. Chemotherapy will be protocol-approved chemotherapy regimen containing intravenous Doxorubicin (or Epirubicin), Cyclophosphamide, and Paclitaxel (or Docetaxel).

Patients receive a protocol-approved chemotherapy regimen containing Doxorubicin (or Epirubicin), Cyclophosphamide, and Paclitaxel (or Docetaxel) based on the patient and/or physician preference.

Mathematical modeling using the patient's diagnostic core biopsy and baseline MRI of the breast will be used to predict the response to above therapy.

Following the completion of neoadjuvant chemotherapy, surgical approach and adjuvant radiation and endocrine therapy are left to the discretion of the treating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Women with newly diagnosed human epidermal growth factor receptor 2 (HER2)-negative, estrogen receptor (ER) positive or negative, progesterone receptor (PR) positive or negative infiltrating ductal carcinoma (IDC) of the breast
* Clinically stage II-III
* Patients with inflammatory, multifocal, multicentric and synchronous bilateral breast cancers are allowed. However, in patients with inflammatory breast cancer, patients must have a measurable, biopsied mass within the breast pre-chemotherapy.
* Willing and able to provide informed consent
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1
* Patients must be able to receive neoadjuvant anthracycline / taxane based chemotherapy in the opinion of the treating physician. Criteria include:

  * Adequate bone marrow function, as defined by peripheral granulocyte count of ≥ 1,500/mm3, and platelet count ≥100,000/mm3
  * Adequate renal function with creatinine levels ≤ 1.5 X the upper limit of normal and estimated glomerular filtration rate (eGFR) >30.
  * Adequate liver function with a bilirubin, Alkaline phosphatase and transaminases (ALT and AST) of ≤ 1.5 X the institutional upper limit of normal.
  * Multigated acquisition (MUGA) or echocardiogram (ECHO) demonstrating a left ventricular ejection fraction (LVEF) within institutional normal limits
* Women of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients may also co-enroll in trials that compare local therapies, or compare systemic adjuvant therapies.
* Patients must have had (or be scheduled to have) a pre neoadjuvant chemotherapy MRI of the breast with gadolinium contrast as part of their planned routine breast cancer care.

Exclusion Criteria:

* Patients must not have had surgery or radiation or begun chemotherapy or endocrine therapy for their breast cancer prior to registration.
* Patients must not be pregnant or nursing due to the possibility of harm to a fetus or nursing infant from this treatment regimen.
* Presence of electrically, magnetically, or mechanically activated implants including cardiac pacemakers, cochlear implants, magnetic surgical clips or prosthesis that would preclude MRI.
* History of severe claustrophobia
* History of allergic reaction to gadolinium
* Patients must not have metastatic disease
* Baseline sensory/motor neuropathy > grade 2
* Clinically significant cardiovascular disease
* Serious intercurrent infection or nonmalignant medical illness
* Creatinine clearance prohibiting the use of gadolinium (eGFR < 30)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with Stage II-III HER2 negative breast cancer who are candidates for neoadjuvant anthracycline / taxane based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of using diagnostic needle core biopsy to mathematically predict ƒkill-path in women with breast cancer undergoing neoadjuvant chemotherapy | 5 years
  To assess the feasibility of using diagnostic needle core biopsy to mathematically predict ƒkill-path (fraction of tumor cells killed calculated using data obtained from histopathology) in 10 women with stage II-III Her2-negative, Estrogen Receptor (ER) positive or negative infiltrating ductal carcinoma (IDC) of the breast undergoing neoadjuvant anthracycline / taxane based chemotherapy.
  Calculation of patient specific distribution of liver portal radii or characteristic vessel radius (rb), BVF, and the distance that drugs diffuse through tumor tissue (L) and ƒkill-path (using the investigators' mathematical model) will be obtained via analysis of pre-chemotherapy hematoxylin and eosin (H and E) stained section of diagnostic needle core biopsy specimen. Feasibility of the primary objective will be claimed if the necessary minimum samples are collected to calculate these parameters in 60% of patients.
Feasibility of calculating tumor BVF from pre-chemotherapy gadolinium enhanced MRI of the breast in women with breast cancer undergoing neoadjuvant chemotherapy | 5 years
  To assess the feasibility of calculating patient specific fraction of blood volume within the tumor (tumor BVF) using data obtained from radiographic imaging (ƒkill-rad) from pre-chemotherapy gadolinium enhanced magnetic resonance imaging (MRI) of the breast in 10 women with stage II-III Her2-negative, ER positive or negative infiltrating ductal carcinoma (IDC) of the breast undergoing neoadjuvant anthracycline / taxane based chemotherapy.
  Calculation of patient specific BVF (using the investigators' mathematical model) will be obtained via analysis of pre-chemotherapy gadolinium enhanced MRI of the breast. Feasibility of the secondary objective will be claimed if the necessary minimum samples are collected to calculate these parameters in 60% of patients.
Feasibility of calculating ƒkill-rad from pre-chemotherapy gadolinium enhanced MRI of the breast in women with breast cancer undergoing neoadjuvant anthracycline / taxane based chemotherapy | 5 years
  To assess the feasibility of calculating patient specific fraction of tumor cells killed using data obtained from radiographic imaging (ƒkill-rad) from pre-chemotherapy gadolinium enhanced magnetic resonance imaging (MRI) of the breast in 10 women with stage II-III Her2-negative, ER positive or negative infiltrating ductal carcinoma (IDC) of the breast undergoing neoadjuvant anthracycline / taxane based chemotherapy.
  Calculation of patient specific ƒkill-rad (using the investigators' mathematical model) will be obtained via analysis of pre-chemotherapy gadolinium enhanced MRI of the breast. Feasibility of the secondary objective will be claimed if the necessary minimum samples are collected to calculate these parameters in 60% of patients.

SECONDARY OUTCOMES:
Association between ƒkill-path and ƒkill-rad as calculated with the investigator's mathematical model and response to neoadjuvant chemotherapy at the time of surgery | 5 years
  To evaluate the association between fraction of tumor cells killed using data obtained from histopathology (ƒkill-path) and ƒkill-rad as calculated with the investigators' mathematical model and response to neoadjuvant chemotherapy at the time of surgery.
  The secondary endpoint for describing the association between ƒkillpath and ƒkill-rad is the Spearman correlation coefficient between the two. Endpoints for describing the association between ƒkill-path or ƒkillrad and response will be the mean (SD) and median (Q1-Q3) of ƒkillpath and ƒkill-rad for responders and non-responders. Response will be defined by 1) complete pathologic response (pCR) within the breast and 2) pCR and/or CPS+ EG score < 2 (3).
Association between ƒkill-path and ƒkill-rad and biomarkers as calculated with a mathematical model | 5 years
  To evaluate the association between ƒkill-path and ƒkill-rad as calculated with the investigators' mathematical model and biomarkers associated with tumor angiogenesis, metabolism, acid-base regulation, stress response and invasion.
  The secondary endpoints for describing the association between ƒkill-path and ƒkill-rad and biomarkers associated with tumor angiogenesis, metabolism, acid-base regulation, stress response and invasion are the Spearman correlation coefficients for continuous biomarker measures, or means (SD) and medians (Q1-Q3) of ƒkill-path and ƒkill-rad by levels of categorical biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Ursa Brown-Glaberman, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No